CLINICAL TRIAL: NCT02349178
Title: Bridging Study: A Phase 2 Study Investigating Clofarabine, Cyclophosphamide and Etoposide for Children, Adolescents, and Young Adults (AYA) With Acute Leukemia and Minimal Residual Disease
Brief Title: Bridging Study to Eliminate Presence of MRD for Acute Leukemia Before HCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Medical College of Wisconsin (Other)
Collaborators: American Family Children's Hospital (Other); Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Michael Burke, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bridging
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Leukemia, Acute Lymphoblastic; Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Clofarabine; Cyclophosphamide; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bridging Arm (Experimental): Days 1-5 Receive 20 mg/m2 IV Clofarabine (CLOLAR) over 2 hours followed by 100 mg/m2 IV Etoposide (VP-16, Etopophos) over 2 hours followed by 300 mg/m2 IV Cyclophosphamide (Cytoxan, CTX) as a 30-60 minute infusion
  Interventions: Drug: Clofarabine; Drug: Cyclophosphamide; Drug: Etoposide

INTERVENTIONS:
Drug: Clofarabine — Days 1-5 receive Clofarabine 20 mg/m2 IV over 2 hours
  Other Names: CLOLAR
Drug: Cyclophosphamide — Days 1-5 receive Cyclophosphamide 300 mg/m2 IV as a 30-60 minute infusion
  Other Names: Cytoxan, CTX
Drug: Etoposide — Days 1-5 receive Etoposide 100 mg/m2 IV over 2 hours
  Other Names: VP-16, Etopophos

SUMMARY:
This is a Phase 2 study designed for the purpose of estimating various parameters surrounding the efficacy of Clofarabine, Cyclophosphamide and Etoposide in eliminating minimal residual disease (MRD) in acute leukemia patients otherwise in remission and without causing significant delay of HCT due to treatment related toxicity.

A single course of "bridge" chemotherapy is given prior to the transplant procedure as an approach to improved disease-free survival in a patient group who historically has had inferior outcomes.

DETAILED DESCRIPTION:
Study entry is open to patients regardless of gender or ethnic background.

The intent of this study design is for all patients to receive and complete one course of therapy. Patients who exhibit signs of disease progression or experience an unacceptable toxicity will be discontinued from treatment.

There will be no dose delays or dose reductions of study drugs for hematologic toxicity during Consolidation "Bridging" therapy (Day 1 through Day 30); however, prolonged hematopoietic recovery or bone marrow aplasia during the first 42 days may meet a study stopping rule.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML) with < 5% blasts in the bone marrow (M1) by morphology and that meets one of the following criteria:

Flow cytometric evidence of MRD (≥ 0.01% leukemic blasts for ALL or ≥ 0.5% leukemic blasts for AML detected in the bone marrow) OR Molecular/cytogenetic evidence of disease (FISH or PCR methodology) performed within 7 days And with the intent of going on to an allogeneic hematopoietic cell transplantation (HCT) independent of this study

* Patients must have an available donor and have intention of proceeding directly to ALL-HCT after completion of 1 cycle of Bridging therapy.
* Age 0 to 39 years
* Karnofsky Performance Status ≥ 50% for patients 16 years and older and Lansky Play Score ≥ 50 for patients under 16 years of age (see Appendix 2)
* Patients must have a life expectancy ≥ 8 weeks as determined by the enrolling investigator
* Have acceptable organ function as defined within 7 days of study registration

Renal: creatinine clearance ≥ 60 mL/min/1.73 m2 or serum creatinine based on age/gender as follows:

Hepatic: ALT < 5 x upper limit of normal (ULN) and total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age Cardiac: left ventricular ejection fraction ≥ 40% by ECHO/MUGA

* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. At least 7 days must have elapsed from prior chemotherapy.
* Hematopoietic Growth Factors: At least 7 days since the completion of therapy with a growth factor and at least 14 days since pegfilgrastim (Neulasta®) administration.
* Sexually active females of child bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment and for 2 months after the last dose of chemotherapy. Sexually active men must agree to use barrier contraceptive for the duration of treatment and for 2 months after the last dose of chemotherapy.
* Voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Acute Promyelocytic Leukemia (APL)
* Active extramedullary disease (CNS ≥ CNS2 and/or testicular leukemia) or presence of chloromatous disease
* Receiving concomitant chemotherapy, radiation therapy; immunotherapy or other anti-cancer therapy other than is specified in the protocol
* Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Pregnant or lactating. The agents used in this study are known to be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.
* Known allergy to any of the agents or their ingredients used in this study
* Participating in a concomitant Phase 1 or 2 study

Max Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Burke, MD, Principal Investigator — Medical College of Wisconsin
Locations (4):
- United States (4):
  - Nationwide Children's Hospital, Columbus, Ohio
  - American Family Children's Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bridging Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bridging Arm
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Minimal Residual Disease
Description: A bone marrow evaluation to determine study response and remission status will be performed on study Day 30 or upon adequate blood count recovery (ANC > 0.50 and platelet > 50,000), whichever occurs first. If the marrow is hypocellular and without evidence of normal tri-lineage hematopoiesis the marrow should be repeated at Day 42.
Time Frame: Day 30 or adequate blood recovery
Measure: Count of Participants; unit: Participants
Arm/Group | Bridging Arm
Number analyzed (Participants) | 6
Participants
  MRD Positive | 3
  MRD Negative | 3

ADVERSE EVENTS:
Time Frame: Up to Day 60 from start of study drug
Arm/Group | Bridging Arm
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bridging Arm (N=6)
acute kidney injury (Renal and urinary disorders) | 1 (1) — Creatinine increased - Patient presented to clinic with elevated creatinine x3 from baseline. Patient admitted for IV fluids and monitoring on 5/18/15. Progressed to acute kidney injury
Sepsis (Infections and infestations) | 1 (1) — Patient presented with a heart rate in the 150s and feeling very weak and with a sore throat. She met the criteria for severe sepsis and was admitted to their intensive care unit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT02349178/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT02349178/ICF_001.pdf